CLINICAL TRIAL: NCT05065489
Title: Self-control, Appetite and Psychotic Diagnose: a Resting State EEG Cross Section Study
Brief Title: Resting State Electroencephalogram for Psychotic Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Other Study IDs: WU2021EEG
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Schizophrenia; Bipolar Disorder; Depression
Keywords: electroencephalography; Eating behavior; self control
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depression; Feeding Behavior; Self-Control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Schizophrenia patients: patients who diagnosed with schizophrenia in accordance with DSM-5 criteria
  Interventions: Other: No intervention
- Bipolar disorder patients: patients who diagnosed with bipolar disorder in accordance with DSM-5 criteria
  Interventions: Other: No intervention
- Depression patients: patients who diagnosed with major depression disorder in accordance with DSM-5 criteria
  Interventions: Other: No intervention
- Health control: health participants who have not diagnosed with any psychological or psychiatric disease.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Electroencephalography (EEG) has been proposed as a neurophysiological biomarker to delineate psychotic disorders. Meanwhile, the increased appetite, which might related to self-control process, has been an increasing concern for the management of psychotic disorders. In this cross-section study, investigators collect the resting state EEG data, self-control related scale, eating behaviour questionnaire and psychotic syndrome related assessement and try to find the connection between those measurers, in order to provide novel understanding on the mechanism of psychotic diseases.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with schizophrenia or bipolar disorder or MDD in accordance with DMS-5 Informed Consent

Exclusion Criteria:

Diagnosed with other mental disease in accordance with DSM-5 Comorbid with other severe physiological disease Drug or alcohol abuse Pregnant or lactating

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants were recuited for single center, second xiangya hospital psychiatry department. Both inpatients and outpatients were recuited.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
resting state EEG | baseline
  resting state electroencephalography

SECONDARY OUTCOMES:
Three factor eating questionnaire | baseline
  min value 21, max value 84. The higher scores mean more unhealthy eating behavior.
Barratt Impulsivity Scale | baseline
  min score 26, max score 104. The higher score means more impulsive.
Self-Control Scale | baseline
  min score 36, max score 180. The higher score means less self control.
The positive and negative syndrome scale | baseline
  min score 30, max score 210. The higher score means more severe symptoms.
Hamilton anxiety rating scale | baseline
  min score 14, max score 56. The higher score means more severe anxiety symptom
Hamilton depression rating scale | baseline
  min score 17, max score 68. The higher score means more severe depressive symptom
Young manic rating scale | baseline
  min score 0, max score 60, the higher score means more severe manic syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute of 2nd Xiangya Hospital,CSU, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No